CLINICAL TRIAL: NCT04319341
Title: Obstetric Antiphospholipid Antibody Syndrome : Contribution of the Evaluation of ADAMTS13 Made at the Diagnosis of Pregnancy on Evaluation the Risk of Pre-eclampsia
Acronym: NOH-ADAMTS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: Local/2020/JCG-01
Record Dates: First submitted 2020-03-19; First posted 2020-03-24 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2021-01

CONDITIONS: Antiphospholipid Antibody Syndrome in Pregnancy
MeSH Terms: interventions — ADAMTS13 Protein; Autoantibodies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: To study the prognostic value on the occurrence of pre-eclampsia, ADAMTS13 (ADAMTS13 protein and autoantibodies) in patients diagnosed with oAPS — ADAMTS13 activity, ADAMS13 antigen and anti-ADAMTS13 autoantibodies: U/ml.

SUMMARY:
Study based on data concerning the first pregnancy treated and followed up after the diagnosis of oAPS in the NOH-APS cohort, according to clinical results already published; and on a thematic library collected and preserved at the time of the positive pregnancy test.

ADAMTS 13 will be explored in the available samples defined above: ADAMTS13 antigen (presence of the molecule), ADAMTS13 activity (VWF proteolysis activity of the molecule), global autoantibodies against ADAMTS13 (plasma antibodies recognizing solid phase insolubilized ADAMTS13), these 3 parameters for the description of ADAMTS13 being measured using commercially available diagnostic kits, ELISA type, Technozyme® range, Technoclone, Vienna, Austria.

The clinical endpoint evaluated will be the occurrence (yes/no) of preeclampsia, which is assessed globally, all subtypes combined. Then evaluated according to subtype: late preeclampsia from 34 weeks, early preeclampsia before 34 weeks, eclampsia (convulsions), HELLP syndrome, preeclampsia associated with the birth of a small-for-gestational-age child (defined at percentile 10 of the tables adjusted for gestational age and sex; severe: defined at percentile 3), preeclampsia associated with a retro-placental hematoma, ...

ELIGIBILITY:
Inclusion Criteria:

* Presence of frozen plasma samples from the positive pregnancy test blood sample.
* Adult patients, included in the NOH-APS cohort, who have successfully initiated a new pregnancy after diagnosis of oAPS.

Exclusion Criteria:

* Absence of frozen plasma sample from the blood sample from the positive pregnancy test.
* Patient who objected to the use of their data.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an initially pure, non-thrombotic oAPS; included in the NOH-APS cohort; having been followed in Nîmes for their first pregnancy following the diagnosis of oAPS; N=513.
Sampling Method: Non-Probability Sample
Enrollment: 513 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
The quantification, in vitro, of the activity of ADAMTS13 | at inclusion (J0)
  ADAMTS13 function, U/ml.
The quantification, in vitro, of ADAMTS13 antigen | at inclusion (J0)
  ADAMTS13 antigen, U/ml.
The quantification, in vitro, of ADAMTS13 autoantibodies | at inclusion (J0)
  ADAMTS13 autoantibodies, U/ml.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nîmes - Hôpital Universitaire Carémea, Nîmes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bitsadze V, Bouvier S, Khizroeva J, Cochery-Nouvellon E, Mercier E, Perez-Martin A, Makatsariya A, Gris JC. Early ADAMTS13 testing associates with pre-eclampsia occurrence in antiphospholipid syndrome. Thromb Res. 2021 Jul;203:101-109. doi: 10.1016/j.thromres.2021.04.021. Epub 2021 Apr 27. PMID 33989981